CLINICAL TRIAL: NCT01699126
Title: The Endothelium Dysfunction in Patients of Obstructive Sleep Apnea Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 98-2167B
Record Dates: First submitted 2012-08-30; First posted 2012-10-03 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Obstructive Sleep Apnea; CPAP; Endothelium dysfunction; Hypertension
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypertension | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CPAP, Hypertension (Experimental): evaluate the effect on FMD, blood pressure and inflammation after CPAP on OSA
  Interventions: Device: CPAP
- CPAP and statin, Hypertension (Active Comparator): evaluate the effect on FMD, blood pressure and inflammation after CPAP plus statin on OSA patients
  Interventions: Device: CPAP; Drug: Statin
- OSA, statin, Hypertension (Active Comparator): evaluate the effect on FMD, blood pressure and inflammation after statin treatment on OSA
  Interventions: Drug: Statin
- Placebo (No Intervention): We will also measure the FMD, blood pressure and inflammation on patients with only life style modification as in all other patients

INTERVENTIONS:
Device: CPAP — Continuous Positive Airway Pressure is the routine treatment of OSA, patients will be randomly assigned into CPAP treatment group
  Arms: CPAP and statin, Hypertension; CPAP, Hypertension
Drug: Statin — Statin is an lipid lowering medication with anti-inflammatory effect.
  Other Names: rosuvastatin
  Arms: CPAP and statin, Hypertension; OSA, statin, Hypertension

SUMMARY:
study Hypothesis: We hypothesize that CPAP could effectively improve the endothelial dysfunction by anti-inflammatory effect in patients of OSA,and compare to the effect of statin.

DETAILED DESCRIPTION:
Obstructive sleep apnea is a prevalent disorder that affect 2-4% adults in general population. Cardiovascular and Neurocognitive complication were the most common and severe consequence noted in patients of OSA. Endothelial dysfunction is the early pathologic changes in the vascular wall that precede to the clinical cardiovascular events. Endothelial dysfunction with the deficit of vascular relaxation will induce the development of hypertension. Endothelial dysfunction predict the occurrence of ischemic heart disease and cardiovascular events as stroke. The development of endothelial dysfunction significantly remark the early sign of the development of cardiovascular diseases.

Inflammation trigger by oxygen radical in the vascular system were the major pathogenesis of the endothelial dysfunction. Intermittent hypoxia in the patients of OSA during repeated apnea at night will increase the oxygen radicals therefore trigger the cascade of inflammation process. The inflammatory process could be mediated by the activation of the transcription factors such as NF-KB, AP-1 or from the pathway of HIF-1 cascade. Inflammatory cytokine such as HsCRP inducted by the activation of NF-KB and AP-1 will induce the interaction of monocytes and lymphocytes to further injury to the endothelium of vascular wall. TGF-B secreted by lymphocyte will create the remodeling by fibroblast which result in the thickening of vascular wall. Another pathway by VEGF, endothelin 1, or other protein modulated by HIF-1 is also proposed directly injure to the endothelium that cause the following cardiovascular events.

CPAP treatment for OSA were shown to lowering the severity of blood pressure and cardiovascular events in some reports. Although the effect for blood pressure lowering is still controversial, Most reports actually showed marginal effect on reducing BP to 2 mmHg by CPAP. There is still part of OSA patients with hypertension not responding to CPAP treatment.Besides of the effect of CPAP treatment, the compliance of CPAP is still a major concerning in the treatment of OSA. 60% of patients were reported to continue used CPAP in the well-supported sleep center in USA. Even the CPAP is covered by reimbursement in USA, the low compliance of CPAP impede the treatment of cardiovascular complication of OSA. To improve the control of the cardiovascular consequence of OSA, a convenient and well-tolerated intervention is mandatory. Statin, a powerful lipid-lowering medication, is found to have a significant anti-inflammatory effect in several reports. Statin is even suggested in the population of normal cholesterol to prevent the development of cardiovascular event. Statins exert cholesterol-independent, anti-inflammatory and immunomodulatory effects. Pleiotropic effects are typically mediated by HMG-CoA reductase inhibition, are dose dependent and occur rapidly after initiation of statin treatment. In order to evaluate and explore a safe and convenient method in the control of the cardiovascular complication of OSA, we conduct this study.

ELIGIBILITY:
Inclusion Criteria:

- 1.OSA with AHI>30 2.Male patients with hypertension 3.LDL over 130 mg/dL without any lipid-lowering drug therapy in recent 6 months 4.Signed inform consent and cooperative

Exclusion Criteria:

- 1.Non-cooperative 2.Can't sign inform consent. 3.Had proven major cardiovascular complication such as AMI, CVA. 4.Major chronic disorders and inflammatory disorders: such as DM, ESRD, COPD or rheumatoid arthritis. 5.Under anti-inflammatory medication: such as aspirin, NSAID, steroids, theophylline etc. 6.Acute of chronic infection 1 weeks between blood drawing period will be discarded 7.Study medication will be discontinued among subjects who develop myopathy (CK ≥10 times ULN and muscle aches or weakness) or a persistent elevation in ALT (≥3 times ULN on 2 consecutive tests).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-05; Primary Completion 2013-02 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Flow-Mediated dilatation test(FMD) | 6 months
  FMD is the most sensitive physical marker of endothelial function, we measure the FMD changes after treatment

SECONDARY OUTCOMES:
Blood pressure | 6 months
  Hypertension is the most common cardiovascular disease and prevalent in general population. Many factors including age, obesity, DM, atherosclerosis, OSA….etc will trigger hypertension and exacerbate disease condition. There are more and more evidences showing that OSA play an independent role in hypertension therapy.OSA with CPAP therapy had been proved to reduce blood pressure in many papers especially in resisted hypertension.
  However, during OSA therapy, we found that not all OSA patients with CPAP therapy will achieve the additional goal of blood pressure reduction. Therefore, we hypothesize that there is responder and non-responder in OSA patients with hypertension to CPAP therapy. To clarify the character of responder of OSA patients with hypertension and further investigate the mechanism between OSA and hypertension, we aim to conduct this study:

OTHER OUTCOMES:
Hs-CRP | 6 months
  Endothelial dysfunction is supposed to be mediated by inflammation process after hypoxia. Hs-CRP is the most sensitive marker to evaluate the inflammation level.
Inflammatory markers | 6 months
  Inflammation after hypoxia is suggested to be the pathogenesis of endothelial dysfunction. We will measure the inflammatory markers after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: WAN-CHING Ho, M.D., Principal Investigator — Taiwan Society of Cardiology
Locations (1):
- Chang Gang Memorial Hospital, Taoyuan District, Taiwan

REFERENCES:
- [Result] Luthje L, Andreas S. Obstructive sleep apnea and coronary artery disease. Sleep Med Rev. 2008 Feb;12(1):19-31. doi: 10.1016/j.smrv.2007.08.002. Epub 2007 Nov 1. PMID 17936040
- [Result] Bradley TD, Floras JS. Obstructive sleep apnoea and its cardiovascular consequences. Lancet. 2009 Jan 3;373(9657):82-93. doi: 10.1016/S0140-6736(08)61622-0. Epub 2008 Dec 26. PMID 19101028
- [Result] Atkeson A, Yeh SY, Malhotra A, Jelic S. Endothelial function in obstructive sleep apnea. Prog Cardiovasc Dis. 2009 Mar-Apr;51(5):351-62. doi: 10.1016/j.pcad.2008.08.002. PMID 19249441
- [Result] Jelic S, Padeletti M, Kawut SM, Higgins C, Canfield SM, Onat D, Colombo PC, Basner RC, Factor P, LeJemtel TH. Inflammation, oxidative stress, and repair capacity of the vascular endothelium in obstructive sleep apnea. Circulation. 2008 Apr 29;117(17):2270-8. doi: 10.1161/CIRCULATIONAHA.107.741512. Epub 2008 Apr 14. PMID 18413499
- [Result] Gozal D, Kheirandish-Gozal L. Cardiovascular morbidity in obstructive sleep apnea: oxidative stress, inflammation, and much more. Am J Respir Crit Care Med. 2008 Feb 15;177(4):369-75. doi: 10.1164/rccm.200608-1190PP. Epub 2007 Nov 1. PMID 17975198
- [Result] Gilmartin GS, Tamisier R, Curley M, Weiss JW. Ventilatory, hemodynamic, sympathetic nervous system, and vascular reactivity changes after recurrent nocturnal sustained hypoxia in humans. Am J Physiol Heart Circ Physiol. 2008 Aug;295(2):H778-85. doi: 10.1152/ajpheart.00653.2007. Epub 2008 Jun 6. PMID 18539753
- [Result] Iturriaga R, Rey S, Del Rio R. Cardiovascular and ventilatory acclimatization induced by chronic intermittent hypoxia: a role for the carotid body in the pathophysiology of sleep apnea. Biol Res. 2005;38(4):335-40. doi: 10.4067/s0716-97602005000400004. PMID 16579514
- [Result] Williams B. The year in hypertension. J Am Coll Cardiol. 2008 May 6;51(18):1803-17. doi: 10.1016/j.jacc.2008.03.010. No abstract available. PMID 18452788
- [Result] Campos-Rodriguez F. Screening for sleep apnea in patients with resistant hypertension. Am J Hypertens. 2008 Jul;21(7):728. doi: 10.1038/ajh.2008.193. No abstract available. PMID 18584016
- [Result] Haentjens P, Van Meerhaeghe A, Moscariello A, De Weerdt S, Poppe K, Dupont A, Velkeniers B. The impact of continuous positive airway pressure on blood pressure in patients with obstructive sleep apnea syndrome: evidence from a meta-analysis of placebo-controlled randomized trials. Arch Intern Med. 2007 Apr 23;167(8):757-64. doi: 10.1001/archinte.167.8.757. PMID 17452537
- [Result] Phillips CL, Yee B, Yang Q, Villaneuva AT, Hedner J, Berend N, Grunstein R. Effects of continuous positive airway pressure treatment and withdrawal in patients with obstructive sleep apnea on arterial stiffness and central BP. Chest. 2008 Jul;134(1):94-100. doi: 10.1378/chest.07-3121. Epub 2008 Mar 17. PMID 18347202